CLINICAL TRIAL: NCT04844762
Title: Addiction and Behavior Related to Menthol Cigarette Substitutes
Acronym: MENTHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: University of Vermont (Other); Brown University (Other); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: OSU-19145; 1R21DA046333-01A1 (NIH)
Record Dates: First submitted 2020-07-02; First posted 2021-04-14 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Smoking (Tobacco) Addiction
Keywords: Menthol cigarettes
MeSH Terms: conditions — Smoking; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- usual brand menthol cigarette (UBMC) (Active Comparator): Study participant's usual brand menthol cigarette
  Interventions: Behavioral: Menthol cigarettes substitutes; Behavioral: Menthol cigarettes substitutes and menthol cigarettes
- menthol roll-your-own cigarette (mRYO) (Active Comparator): Mentholated pipe tobacco in a roll-your-own cigarette tube
  Interventions: Behavioral: Menthol cigarettes substitutes; Behavioral: Usual brand menthol cigarettes and substitutes; Behavioral: Menthol cigarettes substitutes and menthol cigarettes
- menthol filtered little cigar (mFLC) (Active Comparator): The menthol filtered cigar will be Cheyenne (Cheyennecigars.com) Seneca (senecacigars.com)
  Interventions: Behavioral: Menthol cigarettes substitutes; Behavioral: Usual brand menthol cigarettes and substitutes; Behavioral: Menthol cigarettes substitutes and menthol cigarettes
- non-menthol cigarette (nmC) (Active Comparator): The non-menthol cigarette will be Newport non-menthol cigarettes.
  Interventions: Behavioral: Menthol cigarettes substitutes; Behavioral: Usual brand menthol cigarettes and substitutes; Behavioral: Menthol cigarettes substitutes and menthol cigarettes

INTERVENTIONS:
Behavioral: Menthol cigarettes substitutes — In Phase 1, participants will complete 4 smoking sessions using a different product each session to examine each product's abuse liability.
Behavioral: Usual brand menthol cigarettes and substitutes — In Phase 2, to assess uptake, changes in subjective effects, and use over time, participants will select their preferred study product from Phase 1 and be instructed to completely substitute the product for their usual brand menthol cigarette for one week.
  Arms: menthol filtered little cigar (mFLC); menthol roll-your-own cigarette (mRYO); non-menthol cigarette (nmC)
Behavioral: Menthol cigarettes substitutes and menthol cigarettes — In Phase 3, participants will complete a final in-lab visit to assess the substitutability of their preferred product from Phases 1 and 2, under simulated ban conditions using a progressive ratio task.

SUMMARY:
The goal of the proposed study is to examine the abuse liability and substitutability of plausible menthol cigarette alternatives currently on the market, including menthol filtered little cigars (mFLC), menthol roll-your-own (mRYO) pipe tobacco and cigarette tubes, and non-menthol cigarettes (nmC). In addition, the study will elucidate real-time mechanisms including product characteristics and perceived effects associated with greater substitution.

DETAILED DESCRIPTION:
Using an in-laboratory and ad libitum outpatient mixed design, 80 current menthol cigarette smokers will complete a three phase, 3 week study: in Phase 1, utilizing a randomized crossover design, participants will complete 5 smoking sessions, each session smoking a different product examining each participants puff topography while sampling the product, the products' ability to suppress nicotine craving/withdrawal, and the product's demand indices. Products will include participants usual brand menthol cigarette (UBMC) as well as 3 commercially-available alternatives, including an mFLC, a pre-assembled mRYO product (menthol tobacco and non-menthol tube), and an nmC. All sessions will occur following 12 hours of nicotine abstinence and be separated by 48 hours. In Phase 2, participants will select their preferred study product from Phase 1 and be instructed to completely substitute the product for their UBMC for one week. Participants will complete ecological momentary assessments (EMA) during this period to more accurately assess degree of substitution and perceived effects in real time. In Phase 3, participants will complete a final in-lab visit to assess the substitutability of their preferred product, under simulated ban conditions using a progressive ratio task. In all phases, multiple domains of abuse liability will be assessed, including product administration (in-lab puff topography and EMA self-report measures), product liking and craving and withdrawal suppression (in-lab and EMA self-report), and a hypothetical purchase task to simulate demand.

ELIGIBILITY:
Inclusion criteria:

* current menthol cigarette smoker (>90% menthol cigarette use; ≥5 cigarettes per day) for at least the past 6 months.
* between 18-24 (young adult) or 25-50 years old (aged 25+)
* willing to provide informed consent and abstain from all tobacco and nicotine use for at least 12 hours prior to the five lab sessions
* willing to complete one week of EMA
* read and speak English.

Exclusion criteria:

* self-reported diagnosis of lung disease including asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* history of cardiac event or distress within the past 3 months
* currently pregnant, planning to become pregnant, or breastfeeding (will be verified with urine pregnancy test)
* use of other tobacco products (e.g., e-cig, cigar, etc.) >5 days in the past month
* current marijuana use >5 times per month
* any use of other illicit drugs during the last 30 days (verified by urinalysis at initial visit)
* currently engaging in a smoking cessation attempt
* currently using one of the alternative menthol study products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villanti AC, Hinton A, Schulz JA, Erath TG, Mehta T, Reed D, Tidey J, Businelle M, Wagener TL. Substitutability of menthol cigarette alternatives: a clinical trial. Tob Control. 2025 Apr 1;34(2):154-161. doi: 10.1136/tc-2023-058272. PMID 37963771
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes: In phase 1, participants first use their usual brand menthol cigarettes, then they try menthol roll your own, followed by menthol filtered little cigars, and non-menthol cigarettes during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
- UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars: In phase 1, participants first use their usual brand menthol cigarettes, then they try menthol roll your own, followed by non-menthol cigarettes, and menthol filtered little cigars during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
- UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes: In phase 1, participants first use their usual brand menthol cigarettes, then they try menthol filtered little cigars, followed by menthol roll your own, and non-menthol cigarettes during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
- UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own: In phase 1, participants first use their usual brand menthol cigarettes, then they try menthol filtered little cigars, followed by non-menthol cigarettes, and menthol roll your own during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
- UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars: In phase 1, participants first use their usual brand menthol cigarettes, then they try non-menthol cigarettes, followed by menthol roll your own, and menthol filtered little cigars during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
- UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own: In phase 1, participants first use their usual brand menthol cigarettes, then they try non-menthol cigarettes, followed by menthol filtered little cigars, and menthol roll your own during 4 separate lab visits. In phase 2, participants then substituted the product of their choice for their UBMC for 1 week and completed daily diaries. In phase 3, one final lab visit was conducted with the product chosen prior.
Period: Phase 1 First Smoking Session (2 Hrs)
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 17 | 17 | 17 | 18 | 17 | 17
Completed | 17 | 16 | 15 | 17 | 17 | 16
Not Completed | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 1 | 0 | 1
Period: Phase 1 Second Smoking Session (2 Hrs)
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 17 | 16 | 15 | 17 | 17 | 16
Completed | 16 | 14 | 13 | 13 | 15 | 15
Not Completed | 1 | 2 | 2 | 4 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Withdrawal by Study Team | 1 | 2 | 0 | 0 | 0 | 0
Period: Phase 1 Third Smoking Session (2 Hrs)
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 16 | 14 | 13 | 13 | 15 | 15
Completed | 14 | 14 | 13 | 13 | 14 | 15
Not Completed | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Study Team | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Fourth Smoking Session (2 Hrs)
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 14 | 14 | 13 | 13 | 14 | 15
Completed | 13 | 13 | 13 | 13 | 14 | 14
Not Completed | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2 - 1 Week of Daily Diaries
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 13 | 13 | 13 | 13 | 14 | 14
Menthol Roll Your Own | 9 | 9 | 9 | 8 | 7 | 10
Menthol Filtered Little Cigars | 1 | 2 | 1 | 3 | 2 | 1
Non-Menthol Cigarettes | 3 | 2 | 3 | 2 | 5 | 3
Completed | 13 | 13 | 13 | 13 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 3 Chosen Product Visit (~3 Hrs)
Arm/Group | UBMC - Menthol Roll Your Own - Menthol Filtered Little Cigars - Non-menthol Cigarettes | UBMC - Menthol Roll Your Own - Non-menthol Cigarettes - Menthol Filtered Little Cigars | UBMC - Menthol Filtered Little Cigars - Menthol Roll Your Own - Non-menthol Cigarettes | UBMC - Menthol Filtered Little Cigars - Non-menthol Cigarettes - Menthol Roll Your Own | UBMC - Non-menthol Cigarettes - Menthol Roll Your Own - Menthol Filtered Little Cigars | UBMC - Non-menthol Cigarettes - Menthol Filtered Little Cigars - Menthol Roll Your Own
Started | 13 | 13 | 13 | 13 | 14 | 14
Completed | 13 | 13 | 13 | 12 | 14 | 14
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 Participants were enrolled in the study but either withdrew or were lost to follow-up prior to baseline demographic measures being recorded
Groups:
- Overall Population: Full population of participants assessed at baseline.
Arm/Group | Overall Population
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.04 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 68
  More than one race | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 98
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] | 11.90 (5.49)

OUTCOME MEASURES:

1. Primary Outcome: Puffing Topography: Puff Duration
Description: Average puff duration for each participant, in seconds.
Time Frame: Phase 1, Four visits; 20 minute puffing session in total.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
Number analyzed (Puffs) | 991 | 846 | 848 | 832
seconds | 1.99 (0.56) | 2.06 (0.65) | 2.66 (0.95) | 1.87 (0.61)

2. Primary Outcome: Puffing Topography: Inter-puff-interval
Description: Inter-puff-interval, the average time between each puff for each participant, in seconds.
Time Frame: Phase 1, Four visits; 20 minute puffing session in total.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
Number analyzed (Puffs) | 991 | 846 | 848 | 832
seconds | 27.55 (1.73) | 27.54 (1.22) | 26.25 (3.04) | 27.79 (1.61)

3. Primary Outcome: Puffing Topography: Puff Flow Rate
Description: Puff flow rate, the average rate of air flow during each puff for each participant, in ml/second.
Time Frame: Phase 1, Four visits; 20 minute puffing session in total.
Measure: Mean (Standard Deviation); unit: ml/second
Units Other Than Participants: Puffs
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
Number analyzed (Puffs) | 991 | 846 | 848 | 832
ml/second | 23.75 (7.02) | 24.95 (7.66) | 16.97 (5.43) | 22.12 (7.46)

4. Primary Outcome: Puffing Topography: Total Puff Volume
Description: The total volume of all puffs taken for each participant, in ml.
Time Frame: Phase 1, Four visits; 20 minute puffing session in total.
Measure: Mean (Standard Deviation); unit: ml
Units Other Than Participants: Puffs
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
Number analyzed (Puffs) | 991 | 846 | 848 | 832
ml | 462.92 (141.00) | 485.68 (126.65) | 434.66 (127.95) | 391.24 (129.93)

5. Primary Outcome: Drug Effects/Liking Questionnaire
Description: An adapted version of the Drug Effects/Liking Questionnaire will assess the desire and liking of UBMC and all three study products, positive and negative effects (i.e., side effects), and perceived strength and effectiveness. Five visual analog scale items ranging from 0 ('not at all') to 100 ('extremely') assessed wanting to smoke the product again, liking the product, enjoying the product, finding the product pleasurable and satisfying.
Time Frame: Phases 1 and 3 - Up to 3 weeks
Population: In the final in-lab visit (Phase 3) only the participants' preferred product was assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
units on a scale
  Want (Phase 1) | 91.49 (19.09) | 56.68 (29.42) | 26.72 (28.30) | 30.35 (31.74)
  Like (Phase 1) | 96.02 (8.73) | 59.36 (30.89) | 27.93 (28.84) | 30.95 (32.10)
  Enjoy (Phase 1) | 95.02 (11.35) | 57.75 (31.61) | 28.78 (29.31) | 31.58 (32.62)
  Pleasurable (Phase 1) | 94.65 (10.96) | 57.92 (32.79) | 27.65 (29.54) | 32.16 (32.94)
  Satisfying (Phase 1) | 96.09 (8.00) | 60.70 (32.30) | 28.67 (28.49) | 35.17 (33.04)
  Want (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Want (Phase 3) |  | 44.90 (30.52) | 36.80 (38.80) | 44.44 (33.64)
  Like (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Like (Phase 3) |  | 54.39 (32.07) | 52.50 (35.16) | 51.11 (30.12)
  Enjoy (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Enjoy (Phase 3) |  | 53.33 (31.45) | 47.30 (38.39) | 50.44 (30.62)
  Pleasurable (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Pleasurable (Phase 3) |  | 52.18 (32.09) | 44.20 (40.75) | 49.00 (31.52)
  Satisfying (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Satisfying (Phase 3) |  | 57.55 (31.65) | 51.80 (40.56) | 57.06 (29.97)

6. Primary Outcome: Modified Cigarette Evaluation Questionnaire (mCEQ)
Description: The modified Cigarette Evaluation Questionnaire (mCEQ) will assess subjective responses to cigarettes (e.g., reward, satisfaction). The 11-item mCEQ includes five subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction, with items rated from 1 (not at all) to 7 (extremely likely). Items are averaged to create each of the subscales also ranging from 1 to 7 with higher values indicating greater levels of smoking satisfaction, psychological reward, aversion, enjoyment of respiratory tract sensations, an craving reduction.
Time Frame: Phase 1 - Up to 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
score on a scale
  Smoking Satisfaction | 5.79 (1.12) | 4.06 (1.70) | 2.43 (1.32) | 2.59 (1.61)
  Psychological Reward | 3.97 (1.45) | 2.85 (1.49) | 2.03 (1.25) | 2.54 (1.43)
  Aversion | 2.23 (1.04) | 1.98 (1.14) | 1.66 (1.22) | 2.45 (1.29)
  Enjoyment of Respiratory Tract Sensations | 5.18 (1.43) | 3.80 (1.85) | 2.21 (1.50) | 2.59 (1.64)
  Craving Reduction | 5.12 (1.66) | 4.63 (1.70) | 3.02 (1.71) | 3.83 (1.79)

7. Primary Outcome: Modified Cigarette Evaluation Questionnaire (mCEQ)
Description: as for outcome 6
Time Frame: Phase 3 - Approximately 3 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 51 | 10 | 18
score on a scale
  Smoking Satisfaction | 3.89 (1.74) | 3.43 (1.94) | 3.52 (1.83)
  Psychological Reward | 2.90 (1.66) | 2.26 (1.84) | 2.58 (1.38)
  Aversion | 1.62 (1.23) | 1.15 (0.24) | 1.67 (1.22)
  Enjoyment of Respiratory Tract Sensations | 3.63 (1.88) | 2.70 (2.16) | 3.17 (1.69)
  Craving Reduction | 4.31 (1.73) | 3.80 (1.93) | 4.06 (1.76)

8. Primary Outcome: Cigarette Purchase Task
Description: The Cigarette Purchase Task will ask participants how much they would be willing to pay (ranging from 0 cents to $1) to smoke each product. Given that the study products will look similar to cigarettes, we will retain the original language (e.g., 1 cigarette) in the purchase task. Willingness to spend more will indicate greater abuse liability. Pmax (the price associated with the maximal expenditure, i.e., the highest price before the curve changes from inelastic to elastic), and breakpoint (the last price in which consumption is greater than 0) are reported.
Time Frame: Phase 1 - Up to 2 weeks
Measure: Mean (95% Confidence Interval); unit: Dollars
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
Dollars
  Pmax | 2.03 [1.56 to 2.49] | 1.64 [1.23 to 2.05] | 1.63 [0.88 to 2.37] | 1.57 [1.01 to 2.13]
  Breakpoint | 6.12 [4.35 to 7.90] | 4.30 [2.76 to 5.78] | 2.82 [1.53 to 4.11] | 3.15 [1.93 to 4.36]

9. Primary Outcome: Cigarette Purchase Task
Description: as for outcome 8
Time Frame: Phase 3 - Approximately 3 hours
Measure: Mean (95% Confidence Interval); unit: Dollars
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 49 | 9 | 17
Dollars
  Pmax | 1.62 [1.21 to 2.03] | 1.11 [0.03 to 2.20] | 1.03 [0.54 to 1.52]
  Breakpoint | 3.36 [2.18 to 4.55] | 4.51 [-2.95 to 11.97] | 2.69 [1.04 to 4.33]

10. Primary Outcome: Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form (Modified)
Description: Smoking urges/craving will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form. This is a 10-item measure where participants rate smoking-related items (All I want right now is a cigarette) on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 with higher scores indicating greater craving to smoke.
Time Frame: Phase 1-3 - Up to 3 weeks
Population: In phases 2 and 3 only the participants' preferred product was assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
score on a scale
  Desire (0 Minutes; Phase 1) | 30.24 (5.93) | 29.63 (7.04) | 29.77 (7.19) | 29.77 (7.08)
  Desire (5 Minutes; Phase 1) | 12.72 (8.51) | 11.60 (7.38) | 15.16 (8.72) | 11.54 (7.66)
  Desire (15 Minutes; Phase 1) | 14.90 (8.82) | 14.31 (9.02) | 17.71 (9.08) | 14.60 (8.60)
  Desire (30 Minutes; Phase 1) | 17.00 (9.43) | 16.50 (9.24) | 19.96 (9.56) | 17.23 (9.25)
  Desire (60 Minutes; Phase 1) | 19.92 (9.33) | 20.17 (9.41) | 22.38 (9.84) | 20.51 (9.71)
  Desire (90 Minutes; Phase 1) | 22.92 (9.06) | 23.23 (9.22) | 24.85 (9.39) | 23.27 (9.49)
  Relief (0 Minutes; Phase 1) | 18.00 (7.30) | 18.65 (8.99) | 17.84 (8.89) | 18.23 (9.32)
  Relief (5 Minutes; Phase 1) | 8.24 (4.78) | 7.82 (4.66) | 9.48 (5.59) | 7.83 (4.43)
  Relief (15 Minutes; Phase 1) | 8.52 (5.04) | 9.05 (5.46) | 10.78 (6.58) | 9.31 (5.49)
  Relief (30 Minutes; Phase 1) | 9.21 (5.72) | 10.26 (6.05) | 11.89 (6.89) | 10.82 (6.61)
  Relief (60 Minutes; Phase 1) | 10.38 (6.33) | 12.29 (7.41) | 13.05 (7.65) | 12.06 (6.99)
  Relief (90 Minutes; Phase 1) | 11.84 (6.76) | 13.92 (7.90) | 14.39 (7.69) | 13.14 (7.42)
  Desire (Phase 2): number analyzed (Participants) | 0 | 52 | 10 | 18
  Desire (Phase 2) |  | 16.79 (6.70) | 9.87 (4.04) | 13.74 (7.19)
  Relief (Phase 2): number analyzed (Participants) | 0 | 52 | 10 | 18
  Relief (Phase 2) |  | 11.27 (5.75) | 6.94 (2.56) | 9.79 (5.39)
  Desire (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Desire (Phase 3) |  | 9.92 (5.77) | 10.70 (8.71) | 14.11 (10.53)
  Relief (Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  Relief (Phase 3) |  | 7.37 (3.10) | 6.90 (3.28) | 10.22 (8.12)

11. Primary Outcome: Minnesota Nicotine Withdrawal Scale
Description: Nicotine withdrawal will be assessed using the empirically validated 15-item version of the Minnesota Nicotine Withdrawal Scale (MNWS). Items were rated on a 5-point scale from 0 (none) to 4 (severe). This measure assesses smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing). MNWS is the sum of 7 items with scores ranging from 0 to 28 and MNWS Craving is a single item with scores ranging from 0 to 4, higher scores indicate a greater craving.
Time Frame: Phase 1-3 - Up to 3 weeks
Population: In phases 2 and 3 only the participants' preferred product was assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 98 | 84 | 82 | 83
score on a scale
  MNWS (90min, Phase 1) | 4.59 (4.94) | 4.95 (5.44) | 5.17 (5.60) | 4.73 (4.88)
  MNWS Craving (90min, Phase 1) | 2.34 (1.30) | 2.17 (1.40) | 2.40 (1.46) | 2.11 (1.52)
  MNWS (7 day average, Phase 2): number analyzed (Participants) | 0 | 52 | 10 | 18
  MNWS (7 day average, Phase 2) |  | 12.89 (5.55) | 7.88 (1.06) | 12.29 (5.13)
  MNWS (Post PR Task, Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  MNWS (Post PR Task, Phase 3) |  | 3.80 (4.62) | 1.60 (2.27) | 4.83 (5.38)
  MNWS Craving (Post PR Task, Phase 3): number analyzed (Participants) | 0 | 51 | 10 | 18
  MNWS Craving (Post PR Task, Phase 3) |  | 0.59 (0.75) | 0.70 (1.25) | 0.83 (1.15)

12. Primary Outcome: Subjective Effects (EMA)
Description: Subjective effects (EMA) of the Phase 2 substitute product will be derived from daily diary EMAs assessing product satisfaction and pleasure. Self-report measure with items rated from 1 (not at all) to 7 (extremely).
Time Frame: Phase 2 - 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 52 | 10 | 18
score on a scale
  Like | 3.80 (1.64) | 3.21 (1.80) | 3.67 (1.30)
  Pleasurable | 3.70 (1.64) | 2.93 (1.81) | 3.61 (1.31)

13. Primary Outcome: Cross Price Elasticity Task
Description: A Cross-Price Task in Phases 1 and 3 will estimate substitutability of the study product for the UBMC. Participants will be asked how many study products and UBMCs they would consume when the price of the study product is fixed at $1 and the UBMC prices escalate. The data are then fit to an exponential equation that indicates whether the fixed-price product substitutes for the primary product, and the degree of substitution. Cross price elasticity (CPE) for each study product compared to UBMC > 0.2 indicates substitution, CPE < -0.2 indicates complementarity, and CPE between -0.2 and 0.2 indicate independence of the two products.
Time Frame: Phases 1 - Up to 2 weeks
Measure: Mean (95% Confidence Interval); unit: slope
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 49 | 9 | 15
slope | 0.315 [0.235 to 0.396] | 0.085 [0.057 to 0.114] | 0.238 [0.188 to 0.287]

14. Primary Outcome: Cross Price Elasticity Task
Description: as for outcome 13
Time Frame: Phase 3 - Approximately 3 hours
Measure: Mean (95% Confidence Interval); unit: slope
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 49 | 9 | 15
slope | 0.282 [0.203 to 0.360] | 0.216 [0.144 to 0.289] | 0.281 [0.182 to 0.379]

15. Primary Outcome: Progressive Ratio Task (UBMC vs. Study Product)
Description: The PR task will simulate the effect that restricting menthol in cigarettes would have on increasing (or not) preference for other alternative menthol substitutes. Participants will complete a 90-minute concurrent choice task with different cost (effort) required to earn the reinforcement (2 puffs) from their UBMC and the study product (mFLC or mRYO). Puffs from the study product can be earned by clicking a computer mouse 10 times on a picture of the study product, but to earn two puffs of the UBMC, they will required to make escalating response requirements (computer mouse clicks) according to the following schedule: 10, 160, 320, 640, 1280, 2400, 3600, 4800, 6000, 7200, and 8400. A maximum of 10 reinforcers (20 puffs) per session will be allowed. Participants will be informed of the different sequence between products and instructed that the session are 3 hours in length no matter how much or how little they respond.
Time Frame: Phase 3 - Approximately 3 hours
Measure: Mean (Standard Deviation); unit: Number of Puffs on UBMC
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 51 | 10 | 18
Number of Puffs on UBMC | 5.47 (1.75) | 4.70 (2.21) | 5.06 (1.73)

16. Primary Outcome: Use Behavior (EMA)
Description: Participants will receive on EMA delivered randomly during the day and an evening daily diary (around 30mins before bedtime). Random EMAs will assess: mood, affect, nicotine craving and withdrawal symptoms, stress, recency of smoking, alcohol use, current setting, and switching self-efficacy; daily diary EMAs will assess UBMC/study product smoked per day, product satisfaction and pleasure. Substitution assessed via use behavior during Phase 2 will be operationalized as the ratio of study product to UBMC used, with a ratio > 0 indicating any substitution and a ratio > 1 indicating substitution of study product for the UBMC at least 50% of the time.
Time Frame: Phase 2 - 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
Number analyzed (Participants) | 52 | 10 | 18
Participants
  Over 50% Substitution | 44 | 8 | 14
  Less than 50% Substitution | 8 | 2 | 4

ADVERSE EVENTS:
Time Frame: Approximately 1 Month
Description: No difference from clinicaltrials.gov definitions
Arm/Group | Usual Brand Menthol Cigarette (UBMC) | Menthol Roll-your-own Cigarette (mRYO) | Menthol Filtered Little Cigar (mFLC) | Non-menthol Cigarette (nmC)
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/84 | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/84 | 0/82 | 0/83
Other Adverse Events (participants affected / at risk) | 6/98 | 4/84 | 3/82 | 2/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Brand Menthol Cigarette (UBMC) (N=98) | Menthol Roll-your-own Cigarette (mRYO) (N=84) | Menthol Filtered Little Cigar (mFLC) (N=82) | Non-menthol Cigarette (nmC) (N=83)
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Depression - sleeps all day and having weight gain
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Depression, Anxiety, and Obsessive Compulsive Disorder
Surgery/cyst removed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Surgery to remove cyst in right hand
Pulmonary/Upper Respiratory - Smoker's Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Smoker's Cough - gets winded easily and feels like lung capacity is low
Neurology/Confusion/Transient Confusion, disorientation or attention deficit (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ADHD - Attention Deficit Hyperactivity Disorder
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Generalized anxiety and depression
Allergy/Immunology/Autoimmune reaction/Immune System Disorders (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant has chronic fatigue, pain, vertigo, and migraine associated with an autoimmune disorder
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General anxiety
Surgery/Intraoperative Injury/Gallbladder removed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Had gallbladder removed due to having gall stones
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Anxious, impatient, lost, depressed (not diagnosed); feels like this because of husband's health, her job, and her menstrual cycles; has felt this way for years, but more serious now because of husband's surgery; planning to see company counselor
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Feeling depressed
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dizzy brain fog; started after stopped using study product (stopped Sunday; started having symptoms late Monday); unsure of dizzy brain fog cause because she is having trouble wearing a mask (COVID) which makes her dizzy and has been travelling
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Depression and anxiety high; had two deaths in her family on the same day
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Psoriasis flare-up
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Depression due to difficulties with ex-husband
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Feeling moderately depressed; has been taking meds for the last 15 years to control anxiety and depression; has seen doctors and counselors; broke up with her boyfriend and is sad; said depression was not unmanageable
Neurology/Mood alteration/Depression/Mild mood alteration not interfering with function (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Depression because of aunt being in the hospital with COVID

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04844762/Prot_SAP_000.pdf